CLINICAL TRIAL: NCT04693923
Title: Capillary Refill Time Response to a Rapid Fluid Challenge in Septic Shock Patients: Pathophysiological Determinants, and Relation to Changes in Systemic, Regional and Microcirculatory Blood Flow
Brief Title: Capillary Refill Time Response to a Rapid Fluid Challenge in Septic Shock Patients
Acronym: AUSTRALIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Glenn Hernández, Clinical Professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 190527001
Record Dates: First submitted 2020-12-21; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled study in parallel groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (rapid fluid challenge) (Experimental): Patients will receive a rapid fluid challenge (4ml/kg of crystalloids in 5 minutes using a syringe of 60 mL and a timer in the multiparameter monitor).
  Interventions: Procedure: Fluid challenge
- Group B (standard fluid challenge) (Active Comparator): Patients will receive a standard fluid challenge (500 ml of crystalloids in 30 minutes).
  Interventions: Procedure: Fluid challenge

INTERVENTIONS:
Procedure: Fluid challenge — Fluid challenge according to the assigned group

SUMMARY:
In septic shock patients, the hemodynamic coherence between systemic, regional and microcirculatory blood flow can be tracked by "capillary refill time (CRT) response to an increase in stroke volume induced by a rapid fluid challenge". A parallel improvement in regional blood flow, microcirculation and hypoperfusion-related parameters should be expected in CRT-responders as reflection of preserved hemodynamic coherence. CRT non-response is associated with a more severe systemic inflammatory state, endothelial and microvascular dysfunction, and a higher adrenergic tone.

The objective of this study is to determine if CRT response after a rapid fluid challenge signals a state of hemodynamic coherence as demonstrated by a parallel improvement in regional and microcirculatory blood flow in CRT-responders, and to explore the pathophysiological mechanisms associated to CRT non-response.

DETAILED DESCRIPTION:
INTRODUCTION Septic shock is associated with a high mortality risk of up to 30-60%. Multiple pathogenic factors can lead to progressive tissue hypoperfusion in the context of severe systemic inflammation. However, despite extensive research on the best monitoring and resuscitation strategy many uncertainties persist. Over-resuscitation, particularly when inducing fluid overload, might contribute to a worse outcome. Fluid overload more likely occurs when fluids are administered to fluid unresponsive patients, but also when inappropriate resuscitation goals are pursued. The systematic use of bedside techniques to determine fluid responsiveness (FR) can help to avoid fluid overload. Moreover, further deleterious fluid administration can be prevented by adding the evaluation of hemodynamic coherence in parallel or sequentially to FR. Further research on this topic is imperative considering not only the extremely high morbidity and mortality of septic shock, but also the increasing economic burden over the health system in both developed and low/medium income countries.

CAPILLARY REFILL TIME (CRT) AS A TARGET FOR FLUID RESUSCITATION IN SEPTIC SHOCK The skin territory lacks auto-regulatory flow control, and therefore, sympathetic activation impairs skin perfusion during circulatory dysfunction, a phenomenon that can be evaluated by peripheral perfusion assessment. Abnormal peripheral perfusion after initial or advanced resuscitation is associated with increased morbidity and mortality. A cold clammy skin, mottling or prolonged CRT have been suggested as triggers for fluid resuscitation in patients with septic shock. Moreover, the excellent prognosis associated with CRT recovery, its rapid-response time to fluid loading, its relative simplicity, its availability in resource-limited settings, and its capacity to change in parallel with perfusion of physiologically relevant territories such as the hepatosplanchnic region, constitute strong reasons to consider CRT as a target for fluid resuscitation in septic shock patients.

THE CONCEPT OF A FLUID CHALLENGE Since absolute or relative hypovolemia is almost universally present in early septic shock, resuscitation starts with fluid loading in pre-ICU settings. Fluid loading is the rapid administration of fluids without necessarily monitoring the response in real-time, when confronting severe life-threatening hypotension and hypoperfusion. In this setting, usually 20-30 ml/kg crystalloids are loaded.

If circulatory dysfunction is not resolved with this initial management, patients are transferred to the ICU, where advanced fluid resuscitation is started with the fundamental objective to increase systemic blood flow. The initial step is assessment of FR. Fluid-responsive patients will increase stroke volume >10 to 15% after receiving a fluid bolus (usually 250 to 500 ml of crystalloids) since they are in the ascending part of the Starling curve. On the contrary, being fluid-unresponsive implies to be in the flat part of the curve where fluids will only lead to congestion without increasing stroke volume.

The standard practice is to perform a fluid challenge in fluid-responsive patient who are still hypoperfused. A fluid challenge consists of a fluid bolus, large and rapid enough, to increase venous return and cardiac output (CO) in fluid responsive patients, and eventually improve tissue perfusion, depending on the status of hemodynamic coherence (see below). Fluid is given as a fluid challenge so that response can be assessed looking at the target, and the need for ongoing fluid therapy ascertained.

Very few studies have addressed the best way to perform a fluid challenge. A recent study demonstrated that a minimum of 4 ml/kg fluid bolus maximizes the impact on stroke volume. On the other hand, the rate of administration is also important. The FENICE study found that the most common practice in Europe is to administer 500 ml of crystalloids in 30 minutes as a fluid challenge (standard method). However, a more rapid fluid challenge in 5 to 10 minutes might exert more beneficial effects on tissue perfusion by inducing a vasodilatory reflex in addition to the increase in stroke volume. T

THE CONCEPT AND CLINICAL RELEVANCE OF HEMODYNAMIC COHERENCE IN SEPTIC SHOCK Hemodynamic coherence is the condition in which resuscitation of systemic macrohemodynamic variables results in concurrent improvement in regional and microcirculatory flow, and correction of tissue hypoperfusion. Loss of coherence in septic shock is associated with increasing organ dysfunction and a worse prognosis.

The relationship between macrocirculation and regional/microcirculatory blood flow is conditioned by the predominant pathogenic mechanism at different stages of septic shock. At an early stage, hypovolemia and vascular tone depression predominate, leading to low CO and hypotension. An increase in systemic blood flow induced by fluids and/or vasopressors improves regional and microcirculatory flow at this stage. This suggests that macro- and microcirculation are coupled, and should lead to sustained efforts to increase systemic blood flow until hypoperfusion-related variables are corrected.

At a more advanced stage, excessive adrenergic tone (or high-dose vasopressors), and microvascular/endothelial inflammation predominate, leading to abnormal regional flow distribution, and microcirculatory dysfunction that might not respond to systemic blood flow optimization. Microvascular dysfunction occurs because of endothelial dysfunction, leukocyte-endothelium interactions, coagulation and inflammatory disorders, hemorheologic abnormalities, functional shunting, and as an iatrogenic effect of fluid overload/tissue edema.

Hemodynamic coherence is lost in this advanced stage, and efforts to further increase cardiac CO) with fluids or inodilators might lead to fluid overload and the toxicity of vasoactive agents without improving tissue perfusion.

TRACKING THE STATUS OF HEMODYNAMIC COHERENCE IN SEPTIC SHOCK PATIENTS:

A major risk of ICU-based fluid resuscitation is to induce fluid overload. Administering fluids to patients with septic shock after they lost hemodynamic coherence might deteriorate tissue oxygenation, even if they are still fluid-responsive in cardiac function terms. This is a very important consideration. Assessment of hemodynamic coherence is a step forward over the fluid responsiveness concept. This latter looks at the cardiac function curve, but the former instead at the holistic relationship between different components of the cardiovascular system.

The problem is that no single static parameter can predict the status of hemodynamic coherence, and therefore, fluids are abused and probably contribute to progression to refractory shock and death. This is a fundamental contradiction in septic shock resuscitation and highlights the difference between the concepts of FR and hemodynamic coherence. As an example, patients with capillary leak maintain FR along the process because fluids are rapidly lost to the interstitium, and the severe endothelial/microcirculatory dysfunction precludes reperfusion. So, these patients are both fluid-responsive and uncoupled. Moreover, clinicians in despair keep pushing more fluids to try to correct hypoperfusion, which only worsens microcirculatory abnormalities and further impairs perfusion.

Only a novel dynamic test could reveal if the macrocirculation is still coupled or not to regional/microcirculatory blood flow and prevent mismanagement and fluid overload as stated above. The hypothesis of AUSTRALIS is that CRT response to a single rapid fluid challenge can be used as a novel "hemodynamic coherence test." CRT is a sort of bridge between the two worlds (macro-and microcirculation), since it directly represents systemic blood flow (due to the lack of autoregulation), and microcirculation. Normalization of CRT represents an improvement in regional and microcirculatory skin perfusion secondary to an increase in systemic blood flow and/or a reactive decrease in adrenergic tone, thus reflecting hemodynamic coherence. On the contrary, CRT non-response after a rapid fluid challenge is abnormal and a signal of loss of coherence.

PATHOPHYSIOLOGICAL DETERMINANTS OF CRT NON-RESPONSE There are many possible explanations on why CRT might not respond to a stroke volume increase induced by a fluid challenge. Some of these possible mechanisms will be addressed in the proposed study. Adrenergic tone and systemic inflammation, and endothelial/coagulation dysfunction will be addressed by a series of biomarkers selected to provide a broad overview of systemic inflammatory/anti-inflammatory response, and of the transition between endothelial/coagulation activation to established dysfunction, plus direct visualization of microcirculatory status under the tongue, and assessment of microvascular reactivity.

CLINICAL RELEVANCE OF THE PRESENT STUDY If the hypothesis is confirmed, CRT-response to a rapid fluid challenge could be used as a hemodynamic coherence test, and help to avoid futile and dangerous further fluid administration in uncoupled patients, and eventually reduce additional iatrogenic-related excess mortality. Fluid resuscitation could then be focused in fluid responsive patients in whom hemodynamic coherence is still preserved while other perfusion parameters are still not normalized.

Furthermore, establishing the status of hemodynamic coherence with this simple test in pre-ICU or resource-limited settings, could eventually aid in taking triage decisions. CRT non-responders who concentrate septic shock mortality might be rapidly transferred to hospitals with ICU facilities for advanced monitoring and treatment, including reinforcement of source control and eventually rescue therapies.

At the end, this study will help to position CRT, a costless, universally available, and simple test, not only as key target for septic shock resuscitation, but also as a dynamic test of the circulatory function that might help clinicians to interpret the stage of evolution, and help to take timely and critical decisions on fluid resuscitation beyond the concept of fluid responsiveness.

For research purposes, CRT response is defined by "CRT-normalization", and not by "CRT improvement but without normalization" which will be categorized as CRT non-response. This is because hemodynamic tests require to be dichotomous to be applied on a decision branch. In addition, normalization is the only alternative to get certainty that reperfusion has been completed. In any case, partial response will be also included in post-hoc analyses, and the results of the test are not of a binding nature for attending intensivists.

OBJECTIVES AND HYPOTHESIS OR RESEARCH QUESTIONS HYPOTHESIS: In septic shock patients, the hemodynamic coherence between systemic, regional and microcirculatory blood flow can be tracked by "CRT response to an increase in stroke volume induced by a rapid fluid challenge". A parallel improvement in regional blood flow, microcirculation and hypoperfusion-related parameters should be expected in CRT-responders as reflection of preserved hemodynamic coherence. CRT non-response is associated with a more severe systemic inflammatory state, endothelial and microvascular dysfunction, and a higher adrenergic tone.

GENERAL OBJECTIVE: To determine if CRT response after a rapid fluid challenge signals a state of hemodynamic coherence as demonstrated by a parallel improvement in regional and microcirculatory blood flow in CRT-responders, and to explore the pathophysiological mechanisms associated to CRT non-response.

SPECIFIC OBJECTIVES

1. To determine if CRT normalization after an increase in stroke volume (>10%) induced by a rapid fluid challenge is associated with a parallel improvement in regional, microcirculatory blood flow and perfusion variables.
2. To determine if the rate of fluid challenge (rapid vs. standard) influences CRT response rate.
3. To determine if CRT non-response is associated with a more severe systemic inflammatory state, endothelial and microvascular dysfunction, and a higher adrenergic tone.

ELIGIBILITY:
Inclusion Criteria:

1. Septic shock according to the Sepsis-3 Consensus Conference [1], basically septic patients with hypotension requiring norepinephrine (NE) to maintain a MAP of 65 mmHg, and serum lactate levels > 2 mmol/l after initial fluid resuscitation.
2. Less than 24h after fulfilling criteria for septic shock
3. Abnormal CRT (>3 secs)
4. Mechanical ventilation
5. Sinus rhythm with positive predictors of fluid responsiveness [4]
6. Continuous CO monitor, arterial line and central venous catheters in place
7. Required fluid challenge as decided by the attending physician.

Exclusion Criteria:

1. Pregnancy
2. Emergency surgery or dialytic procedure scheduled within the next two hours
3. Do-not-resuscitate status
4. Active bleeding
5. Severe acute respiratory distress syndrome
6. Right ventricular failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Normalization of capillary refill time (CRT) | At baseline, and immediately after the single fluid challenge; then at 30 minutes, and 1, 2, 6 and 24h.
  CRT-response is defined as normalization of the variable after the fluid challenge (normal value CRT ≤3.0 secs).

SECONDARY OUTCOMES:
Procalcitonin | Baseline, and at 6 and 24h after the single fluid challenge
  Inflammation biomarker assessed in serum samples (upper normal limits according to assay)
IL-6 | Baseline, and at 6 and 24h after the single fluid challenge
  Inflammation biomarker assessed in serum samples (upper normal limits according to assay)
IL-10 | Baseline, and at 6 and 24h after the single fluid challenge
  Inflammation biomarker assessed in serum samples (upper normal limits according to assay)
TNF-alpha | Baseline, and at 6 and 24h after the single fluid challenge
  Inflammation biomarker assessed in serum samples (upper normal limits according to assay)
Syndecan-1 | Baseline, and at 6 and 24h after the single fluid challenge
  Marker of endothelial dysfunction, assessed in serum samples (upper normal limits according to assay)
s- ICAM-1 | Baseline, and at 6 and 24h after the single fluid challenge
  Marker of endothelial dysfunction, assessed in serum samples (upper normal limits according to assay)
E-selectin | Baseline, and at 6 and 24h after the single fluid challenge
  Marker of endothelial dysfunction, assessed in serum samples (upper normal limits according to assay)
von Willebrand factor | Baseline, and at 6 and 24h after the single fluid challenge
  Marker of endothelial dysfunction, assessed in serum samples (upper normal limits according to assay)
Platelet count | Baseline, and at 6 and 24h after the single fluid challenge
  Marker of coagulation abnormalities, assessed in serum samples (normal >150.000)
P-selectin | Baseline, and at 6 and 24h after the single fluid challenge
  Marker of coagulation abnormalities, assessed in serum samples (upper normal limits according to assay)
D-Dimer | Baseline, and at 6 and 24h after the single fluid challenge
  Marker of coagulation abnormalities, assessed in serum samples (upper normal limits according to assay)

OTHER OUTCOMES:
Vascular occlusion test assessed by NIRS | Baseline, at 30 min, and at 1, 6 and 24h after the single fluid challenge
  Marker of Microvascular reactivity, assessed by dedicated software
Vascular occlusion test assessed by Laser-Doppler | Baseline, at 30 min, and at 1, 6 and 24h after the single fluid challenge
  Marker of Microvascular reactivity, assessed by dedicated software
Test of thermal challenge with Laser-Doppler, assessed by dedicated software | Baseline, at 30 min, and at 1, 6 and 24h after the single fluid challenge
  Marker of Microvascular reactivity
Epinephrine serial serum levels | Baseline, immediately after, and at 5, at 30 min, and at 1 hour after a single fluid challenge
  Marker of Adrenergic tone, assessed in serum samples (upper normal limits according to assay)
Kidney: renal resistive index | Baseline, and at 5, 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of regional blood flow, assessed by point-of-care ulltrasound
Liver: Indocyanine green plasma disappearance rate | Baseline, at 30 min, and at 1h after a single fluid challenge
  Marker of regional blood flow, assessed with LiMON technique (normal 18-25%)
Muscle tissue oxygenation | Baseline, and at 5, 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of regional blood flow, assessed with NIRS (normal>70%)
Skin blood flow | Baseline, and at 5, 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of regional blood flow, assessed with Laser-Doppler
Sublingual microcirculatory flow and density | Baseline, and at 5, 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of microcirculatory status, assessed with intravital videomicroscopy (PPV<80%, MFI>2.5)
Lactate | Baseline, and at 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of perfusion (normal value <2 mmol/l
ScvO2 | Baseline, and at 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of perfusion (normal value >70%)
pCO2 gradient | Baseline, and at 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of perfusion (normal value <6)
Central venous-arterial pCO2 to arterial-venous O2 content difference ratio | Baseline, and at 30 min, and at 1, 6 and 24h after a single fluid challenge
  Marker of perfusion (normal value <1.4)

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Will be available on a website 6 months after completing recruitment
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after completing recruitment
Access Criteria: Formal request from investigators

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Hernandez G, Bruhn A, Castro R, Regueira T. The holistic view on perfusion monitoring in septic shock. Curr Opin Crit Care. 2012 Jun;18(3):280-6. doi: 10.1097/MCC.0b013e3283532c08. PMID 22473257
- [Background] Malbrain ML, Marik PE, Witters I, Cordemans C, Kirkpatrick AW, Roberts DJ, Van Regenmortel N. Fluid overload, de-resuscitation, and outcomes in critically ill or injured patients: a systematic review with suggestions for clinical practice. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):361-80. doi: 10.5603/AIT.2014.0060. PMID 25432556
- [Background] Jozwiak M, Monnet X, Teboul JL. Prediction of fluid responsiveness in ventilated patients. Ann Transl Med. 2018 Sep;6(18):352. doi: 10.21037/atm.2018.05.03. PMID 30370279
- [Background] Ince C. Hemodynamic coherence and the rationale for monitoring the microcirculation. Crit Care. 2015;19 Suppl 3(Suppl 3):S8. doi: 10.1186/cc14726. Epub 2015 Dec 18. PMID 26729241
- [Background] Machado FR, Cavalcanti AB, Bozza FA, Ferreira EM, Angotti Carrara FS, Sousa JL, Caixeta N, Salomao R, Angus DC, Pontes Azevedo LC; SPREAD Investigators; Latin American Sepsis Institute Network. The epidemiology of sepsis in Brazilian intensive care units (the Sepsis PREvalence Assessment Database, SPREAD): an observational study. Lancet Infect Dis. 2017 Nov;17(11):1180-1189. doi: 10.1016/S1473-3099(17)30322-5. Epub 2017 Aug 17. PMID 28826588
- [Background] Hernandez G, Castro R, Romero C, de la Hoz C, Angulo D, Aranguiz I, Larrondo J, Bujes A, Bruhn A. Persistent sepsis-induced hypotension without hyperlactatemia: is it really septic shock? J Crit Care. 2011 Aug;26(4):435.e9-14. doi: 10.1016/j.jcrc.2010.09.007. Epub 2010 Dec 3. PMID 21126850
- [Background] Hernandez G, Luengo C, Bruhn A, Kattan E, Friedman G, Ospina-Tascon GA, Fuentealba A, Castro R, Regueira T, Romero C, Ince C, Bakker J. When to stop septic shock resuscitation: clues from a dynamic perfusion monitoring. Ann Intensive Care. 2014 Oct 11;4:30. doi: 10.1186/s13613-014-0030-z. eCollection 2014. PMID 25593746
- [Background] Ospina-Tascon GA, Umana M, Bermudez W, Bautista-Rincon DF, Hernandez G, Bruhn A, Granados M, Salazar B, Arango-Davila C, De Backer D. Combination of arterial lactate levels and venous-arterial CO2 to arterial-venous O 2 content difference ratio as markers of resuscitation in patients with septic shock. Intensive Care Med. 2015 May;41(5):796-805. doi: 10.1007/s00134-015-3720-6. Epub 2015 Mar 20. PMID 25792204
- [Background] Tapia P, Soto D, Bruhn A, Alegria L, Jarufe N, Luengo C, Kattan E, Regueira T, Meissner A, Menchaca R, Vives MI, Echeverria N, Ospina-Tascon G, Bakker J, Hernandez G. Impairment of exogenous lactate clearance in experimental hyperdynamic septic shock is not related to total liver hypoperfusion. Crit Care. 2015 Apr 22;19(1):188. doi: 10.1186/s13054-015-0928-3. PMID 25898244
- [Background] Hernandez G, Regueira T, Bruhn A, Castro R, Rovegno M, Fuentealba A, Veas E, Berrutti D, Florez J, Kattan E, Martin C, Ince C. Relationship of systemic, hepatosplanchnic, and microcirculatory perfusion parameters with 6-hour lactate clearance in hyperdynamic septic shock patients: an acute, clinical-physiological, pilot study. Ann Intensive Care. 2012 Oct 15;2(1):44. doi: 10.1186/2110-5820-2-44. PMID 23067578
- [Background] Hernandez G, Boerma EC, Dubin A, Bruhn A, Koopmans M, Edul VK, Ruiz C, Castro R, Pozo MO, Pedreros C, Veas E, Fuentealba A, Kattan E, Rovegno M, Ince C. Severe abnormalities in microvascular perfused vessel density are associated to organ dysfunctions and mortality and can be predicted by hyperlactatemia and norepinephrine requirements in septic shock patients. J Crit Care. 2013 Aug;28(4):538.e9-14. doi: 10.1016/j.jcrc.2012.11.022. Epub 2013 Apr 6. PMID 23566729
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Hernandez G, Tapia P, Alegria L, Soto D, Luengo C, Gomez J, Jarufe N, Achurra P, Rebolledo R, Bruhn A, Castro R, Kattan E, Ospina-Tascon G, Bakker J. Effects of dexmedetomidine and esmolol on systemic hemodynamics and exogenous lactate clearance in early experimental septic shock. Crit Care. 2016 Aug 2;20(1):234. doi: 10.1186/s13054-016-1419-x. PMID 27480413
- [Background] Hernandez G, Bruhn A, Castro R, Pedreros C, Rovegno M, Kattan E, Veas E, Fuentealba A, Regueira T, Ruiz C, Ince C. Persistent Sepsis-Induced Hypotension without Hyperlactatemia: A Distinct Clinical and Physiological Profile within the Spectrum of Septic Shock. Crit Care Res Pract. 2012;2012:536852. doi: 10.1155/2012/536852. Epub 2012 Apr 18. PMID 22570774
- [Background] Cornejo R, Downey P, Castro R, Romero C, Regueira T, Vega J, Castillo L, Andresen M, Dougnac A, Bugedo G, Hernandez G. High-volume hemofiltration as salvage therapy in severe hyperdynamic septic shock. Intensive Care Med. 2006 May;32(5):713-22. doi: 10.1007/s00134-006-0118-5. Epub 2006 Mar 21. PMID 16550372
- [Background] Castro R, Regueira T, Aguirre ML, Llanos OP, Bruhn A, Bugedo G, Dougnac A, Castillo L, Andresen M, Hernandez G. An evidence-based resuscitation algorithm applied from the emergency room to the ICU improves survival of severe septic shock. Minerva Anestesiol. 2008 Jun;74(6):223-31. Epub 2008 Mar 21. PMID 18356807
- [Background] Hernandez G, Pedreros C, Veas E, Bruhn A, Romero C, Rovegno M, Neira R, Bravo S, Castro R, Kattan E, Ince C. Evolution of peripheral vs metabolic perfusion parameters during septic shock resuscitation. A clinical-physiologic study. J Crit Care. 2012 Jun;27(3):283-8. doi: 10.1016/j.jcrc.2011.05.024. Epub 2011 Jul 27. PMID 21798706
- [Background] Lara B, Enberg L, Ortega M, Leon P, Kripper C, Aguilera P, Kattan E, Castro R, Bakker J, Hernandez G. Capillary refill time during fluid resuscitation in patients with sepsis-related hyperlactatemia at the emergency department is related to mortality. PLoS One. 2017 Nov 27;12(11):e0188548. doi: 10.1371/journal.pone.0188548. eCollection 2017. PMID 29176794
- [Background] Hernandez G, Pena H, Cornejo R, Rovegno M, Retamal J, Navarro JL, Aranguiz I, Castro R, Bruhn A. Impact of emergency intubation on central venous oxygen saturation in critically ill patients: a multicenter observational study. Crit Care. 2009;13(3):R63. doi: 10.1186/cc7802. Epub 2009 May 4. PMID 19413905
- [Background] Ospina-Tascon GA, Bautista-Rincon DF, Umana M, Tafur JD, Gutierrez A, Garcia AF, Bermudez W, Granados M, Arango-Davila C, Hernandez G. Persistently high venous-to-arterial carbon dioxide differences during early resuscitation are associated with poor outcomes in septic shock. Crit Care. 2013 Dec 13;17(6):R294. doi: 10.1186/cc13160. PMID 24330804
- [Background] Ospina-Tascon GA, Umana M, Bermudez WF, Bautista-Rincon DF, Valencia JD, Madrinan HJ, Hernandez G, Bruhn A, Arango-Davila C, De Backer D. Can venous-to-arterial carbon dioxide differences reflect microcirculatory alterations in patients with septic shock? Intensive Care Med. 2016 Feb;42(2):211-21. doi: 10.1007/s00134-015-4133-2. Epub 2015 Nov 17. PMID 26578172
- [Background] Palizas F, Dubin A, Regueira T, Bruhn A, Knobel E, Lazzeri S, Baredes N, Hernandez G. Gastric tonometry versus cardiac index as resuscitation goals in septic shock: a multicenter, randomized, controlled trial. Crit Care. 2009;13(2):R44. doi: 10.1186/cc7767. Epub 2009 Mar 31. PMID 19335912
- [Background] Hernandez G, Bruhn A, Luengo C, Regueira T, Kattan E, Fuentealba A, Florez J, Castro R, Aquevedo A, Pairumani R, McNab P, Ince C. Effects of dobutamine on systemic, regional and microcirculatory perfusion parameters in septic shock: a randomized, placebo-controlled, double-blind, crossover study. Intensive Care Med. 2013 Aug;39(8):1435-43. doi: 10.1007/s00134-013-2982-0. Epub 2013 Jun 6. PMID 23740284
- [Background] Regueira T, Bruhn A, Hasbun P, Aguirre M, Romero C, Llanos O, Castro R, Bugedo G, Hernandez G. Intra-abdominal hypertension: incidence and association with organ dysfunction during early septic shock. J Crit Care. 2008 Dec;23(4):461-7. doi: 10.1016/j.jcrc.2007.12.013. Epub 2008 Apr 18. PMID 19056007
- [Background] Hernandez G, Bruhn A, Ince C. Microcirculation in sepsis: new perspectives. Curr Vasc Pharmacol. 2013 Mar 1;11(2):161-9. PMID 23506495
- [Background] Vellinga NA, Boerma EC, Koopmans M, Donati A, Dubin A, Shapiro NI, Pearse RM, Machado FR, Fries M, Akarsu-Ayazoglu T, Pranskunas A, Hollenberg S, Balestra G, van Iterson M, van der Voort PH, Sadaka F, Minto G, Aypar U, Hurtado FJ, Martinelli G, Payen D, van Haren F, Holley A, Pattnaik R, Gomez H, Mehta RL, Rodriguez AH, Ruiz C, Canales HS, Duranteau J, Spronk PE, Jhanji S, Hubble S, Chierego M, Jung C, Martin D, Sorbara C, Tijssen JG, Bakker J, Ince C; microSOAP Study Group. International study on microcirculatory shock occurrence in acutely ill patients. Crit Care Med. 2015 Jan;43(1):48-56. doi: 10.1097/CCM.0000000000000553. PMID 25126880
- [Background] Vellinga NAR, Boerma EC, Koopmans M, Donati A, Dubin A, Shapiro NI, Pearse RM, van der Voort PHJ, Dondorp AM, Bafi T, Fries M, Akarsu-Ayazoglu T, Pranskunas A, Hollenberg S, Balestra G, van Iterson M, Sadaka F, Minto G, Aypar U, Hurtado FJ, Martinelli G, Payen D, van Haren F, Holley A, Gomez H, Mehta RL, Rodriguez AH, Ruiz C, Canales HS, Duranteau J, Spronk PE, Jhanji S, Hubble S, Chierego M, Jung C, Martin D, Sorbara C, Bakker J, Ince C; microSOAP study group. Mildly elevated lactate levels are associated with microcirculatory flow abnormalities and increased mortality: a microSOAP post hoc analysis. Crit Care. 2017 Oct 18;21(1):255. doi: 10.1186/s13054-017-1842-7. PMID 29047411
- [Background] Ince C, Boerma EC, Cecconi M, De Backer D, Shapiro NI, Duranteau J, Pinsky MR, Artigas A, Teboul JL, Reiss IKM, Aldecoa C, Hutchings SD, Donati A, Maggiorini M, Taccone FS, Hernandez G, Payen D, Tibboel D, Martin DS, Zarbock A, Monnet X, Dubin A, Bakker J, Vincent JL, Scheeren TWL; Cardiovascular Dynamics Section of the ESICM. Second consensus on the assessment of sublingual microcirculation in critically ill patients: results from a task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2018 Mar;44(3):281-299. doi: 10.1007/s00134-018-5070-7. Epub 2018 Feb 6. PMID 29411044
- [Background] Ruiz C, Hernandez G, Godoy C, Downey P, Andresen M, Bruhn A. Sublingual microcirculatory changes during high-volume hemofiltration in hyperdynamic septic shock patients. Crit Care. 2010;14(5):R170. doi: 10.1186/cc9271. Epub 2010 Sep 27. PMID 20875109
- [Background] Alegria L, Vera M, Dreyse J, Castro R, Carpio D, Henriquez C, Gajardo D, Bravo S, Araneda F, Kattan E, Torres P, Ospina-Tascon G, Teboul JL, Bakker J, Hernandez G. A hypoperfusion context may aid to interpret hyperlactatemia in sepsis-3 septic shock patients: a proof-of-concept study. Ann Intensive Care. 2017 Dec;7(1):29. doi: 10.1186/s13613-017-0253-x. Epub 2017 Mar 9. PMID 28281216
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Hernandez G, Bellomo R, Bakker J. The ten pitfalls of lactate clearance in sepsis. Intensive Care Med. 2019 Jan;45(1):82-85. doi: 10.1007/s00134-018-5213-x. Epub 2018 May 12. No abstract available. PMID 29754310
- [Background] Hernandez G, Teboul JL. Fourth Surviving Sepsis Campaign's hemodynamic recommendations: a step forward or a return to chaos? Crit Care. 2017 May 30;21(1):133. doi: 10.1186/s13054-017-1708-z. No abstract available. PMID 28592302
- [Background] Bakker J, de Backer D, Hernandez G. Lactate-guided resuscitation saves lives: we are not sure. Intensive Care Med. 2016 Mar;42(3):472-474. doi: 10.1007/s00134-016-4220-z. Epub 2016 Feb 1. No abstract available. PMID 26831675
- [Background] Angus DC. How Best to Resuscitate Patients With Septic Shock? JAMA. 2019 Feb 19;321(7):647-648. doi: 10.1001/jama.2019.0070. No abstract available. PMID 30772916
- [Background] Dubin A, Henriquez E, Hernandez G. Monitoring peripheral perfusion and microcirculation. Curr Opin Crit Care. 2018 Jun;24(3):173-180. doi: 10.1097/MCC.0000000000000495. PMID 29553951
- [Background] Lima A, Bakker J. Clinical assessment of peripheral circulation. Curr Opin Crit Care. 2015 Jun;21(3):226-31. doi: 10.1097/MCC.0000000000000194. PMID 25827585
- [Background] Lima A, Jansen TC, van Bommel J, Ince C, Bakker J. The prognostic value of the subjective assessment of peripheral perfusion in critically ill patients. Crit Care Med. 2009 Mar;37(3):934-8. doi: 10.1097/CCM.0b013e31819869db. PMID 19237899
- [Background] Dumas G, Lavillegrand JR, Joffre J, Bige N, de-Moura EB, Baudel JL, Chevret S, Guidet B, Maury E, Amorim F, Ait-Oufella H. Mottling score is a strong predictor of 14-day mortality in septic patients whatever vasopressor doses and other tissue perfusion parameters. Crit Care. 2019 Jun 10;23(1):211. doi: 10.1186/s13054-019-2496-4. PMID 31182133
- [Background] Coudroy R, Jamet A, Frat JP, Veinstein A, Chatellier D, Goudet V, Cabasson S, Thille AW, Robert R. Incidence and impact of skin mottling over the knee and its duration on outcome in critically ill patients. Intensive Care Med. 2015 Mar;41(3):452-9. doi: 10.1007/s00134-014-3600-5. Epub 2014 Dec 17. PMID 25516087
- [Background] Ait-Oufella H, Bige N, Boelle PY, Pichereau C, Alves M, Bertinchamp R, Baudel JL, Galbois A, Maury E, Guidet B. Capillary refill time exploration during septic shock. Intensive Care Med. 2014 Jul;40(7):958-64. doi: 10.1007/s00134-014-3326-4. Epub 2014 May 9. PMID 24811942
- [Background] Brunauer A, Kokofer A, Bataar O, Gradwohl-Matis I, Dankl D, Bakker J, Dunser MW. Changes in peripheral perfusion relate to visceral organ perfusion in early septic shock: A pilot study. J Crit Care. 2016 Oct;35:105-9. doi: 10.1016/j.jcrc.2016.05.007. Epub 2016 May 12. PMID 27481743
- [Background] van Genderen ME, Engels N, van der Valk RJ, Lima A, Klijn E, Bakker J, van Bommel J. Early peripheral perfusion-guided fluid therapy in patients with septic shock. Am J Respir Crit Care Med. 2015 Feb 15;191(4):477-80. doi: 10.1164/rccm.201408-1575LE. No abstract available. PMID 25679107
- [Background] Ait-Oufella H, Bakker J. Understanding clinical signs of poor tissue perfusion during septic shock. Intensive Care Med. 2016 Dec;42(12):2070-2072. doi: 10.1007/s00134-016-4250-6. Epub 2016 Feb 4. No abstract available. PMID 26846520
- [Background] Cecconi M, Hernandez G, Dunser M, Antonelli M, Baker T, Bakker J, Duranteau J, Einav S, Groeneveld ABJ, Harris T, Jog S, Machado FR, Mer M, Monge Garcia MI, Myatra SN, Perner A, Teboul JL, Vincent JL, De Backer D. Fluid administration for acute circulatory dysfunction using basic monitoring: narrative review and expert panel recommendations from an ESICM task force. Intensive Care Med. 2019 Jan;45(1):21-32. doi: 10.1007/s00134-018-5415-2. Epub 2018 Nov 19. PMID 30456467
- [Background] Cecconi M, Parsons AK, Rhodes A. What is a fluid challenge? Curr Opin Crit Care. 2011 Jun;17(3):290-5. doi: 10.1097/MCC.0b013e32834699cd. PMID 21508838
- [Background] Cecconi M, Hofer C, Teboul JL, Pettila V, Wilkman E, Molnar Z, Della Rocca G, Aldecoa C, Artigas A, Jog S, Sander M, Spies C, Lefrant JY, De Backer D; FENICE Investigators; ESICM Trial Group. Fluid challenges in intensive care: the FENICE study: A global inception cohort study. Intensive Care Med. 2015 Sep;41(9):1529-37. doi: 10.1007/s00134-015-3850-x. Epub 2015 Jul 11. PMID 26162676
- [Background] Carsetti A, Cecconi M, Rhodes A. Fluid bolus therapy: monitoring and predicting fluid responsiveness. Curr Opin Crit Care. 2015 Oct;21(5):388-94. doi: 10.1097/MCC.0000000000000240. PMID 26348418
- [Background] Aya HD, Rhodes A, Chis Ster I, Fletcher N, Grounds RM, Cecconi M. Hemodynamic Effect of Different Doses of Fluids for a Fluid Challenge: A Quasi-Randomized Controlled Study. Crit Care Med. 2017 Feb;45(2):e161-e168. doi: 10.1097/CCM.0000000000002067. PMID 27655325
- [Background] Monge Garcia MI, Guijo Gonzalez P, Gracia Romero M, Gil Cano A, Oscier C, Rhodes A, Grounds RM, Cecconi M. Effects of fluid administration on arterial load in septic shock patients. Intensive Care Med. 2015 Jul;41(7):1247-55. doi: 10.1007/s00134-015-3898-7. Epub 2015 Jun 11. PMID 26077088
- [Background] Roger C, Zieleskiewicz L, Demattei C, Lakhal K, Piton G, Louart B, Constantin JM, Chabanne R, Faure JS, Mahjoub Y, Desmeulles I, Quintard H, Lefrant JY, Muller L; AzuRea Group. Time course of fluid responsiveness in sepsis: the fluid challenge revisiting (FCREV) study. Crit Care. 2019 May 16;23(1):179. doi: 10.1186/s13054-019-2448-z. PMID 31097012
- [Background] Pouska J, Tegl V, Astapenko D, Cerny V, Lehmann C, Benes J. Impact of Intravenous Fluid Challenge Infusion Time on Macrocirculation and Endothelial Glycocalyx in Surgical and Critically Ill Patients. Biomed Res Int. 2018 Nov 1;2018:8925345. doi: 10.1155/2018/8925345. eCollection 2018. PMID 30519590
- [Background] Hoste EA, Maitland K, Brudney CS, Mehta R, Vincent JL, Yates D, Kellum JA, Mythen MG, Shaw AD; ADQI XII Investigators Group. Four phases of intravenous fluid therapy: a conceptual model. Br J Anaesth. 2014 Nov;113(5):740-7. doi: 10.1093/bja/aeu300. Epub 2014 Sep 9. PMID 25204700
- [Background] Edul VS, Enrico C, Laviolle B, Vazquez AR, Ince C, Dubin A. Quantitative assessment of the microcirculation in healthy volunteers and in patients with septic shock. Crit Care Med. 2012 May;40(5):1443-8. doi: 10.1097/CCM.0b013e31823dae59. PMID 22430243
- [Background] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Background] Trzeciak S, McCoy JV, Phillip Dellinger R, Arnold RC, Rizzuto M, Abate NL, Shapiro NI, Parrillo JE, Hollenberg SM; Microcirculatory Alterations in Resuscitation and Shock (MARS) investigators. Early increases in microcirculatory perfusion during protocol-directed resuscitation are associated with reduced multi-organ failure at 24 h in patients with sepsis. Intensive Care Med. 2008 Dec;34(12):2210-7. doi: 10.1007/s00134-008-1193-6. Epub 2008 Jul 2. PMID 18594793
- [Background] Arnemann P, Seidel L, Ertmer C. Haemodynamic coherence - The relevance of fluid therapy. Best Pract Res Clin Anaesthesiol. 2016 Dec;30(4):419-427. doi: 10.1016/j.bpa.2016.11.003. Epub 2016 Nov 10. PMID 27931645
- [Background] Bakker J. Lactate levels and hemodynamic coherence in acute circulatory failure. Best Pract Res Clin Anaesthesiol. 2016 Dec;30(4):523-530. doi: 10.1016/j.bpa.2016.11.001. Epub 2016 Nov 10. PMID 27931655
- [Background] Morelli A, Passariello M. Hemodynamic coherence in sepsis. Best Pract Res Clin Anaesthesiol. 2016 Dec;30(4):453-463. doi: 10.1016/j.bpa.2016.10.009. Epub 2016 Nov 5. PMID 27931649
- [Background] Ospina-Tascon G, Neves AP, Occhipinti G, Donadello K, Buchele G, Simion D, Chierego ML, Silva TO, Fonseca A, Vincent JL, De Backer D. Effects of fluids on microvascular perfusion in patients with severe sepsis. Intensive Care Med. 2010 Jun;36(6):949-55. doi: 10.1007/s00134-010-1843-3. Epub 2010 Mar 11. PMID 20221744
- [Background] Seymour CW, Kennedy JN, Wang S, Chang CH, Elliott CF, Xu Z, Berry S, Clermont G, Cooper G, Gomez H, Huang DT, Kellum JA, Mi Q, Opal SM, Talisa V, van der Poll T, Visweswaran S, Vodovotz Y, Weiss JC, Yealy DM, Yende S, Angus DC. Derivation, Validation, and Potential Treatment Implications of Novel Clinical Phenotypes for Sepsis. JAMA. 2019 May 28;321(20):2003-2017. doi: 10.1001/jama.2019.5791. PMID 31104070
- [Background] Prucha M, Zazula R, Russwurm S. Immunotherapy of Sepsis: Blind Alley or Call for Personalized Assessment? Arch Immunol Ther Exp (Warsz). 2017 Feb;65(1):37-49. doi: 10.1007/s00005-016-0415-9. Epub 2016 Aug 24. PMID 27554587
- [Background] Nesseler N, Martin-Chouly C, Perrichet H, Ross JT, Rousseau C, Sinha P, Isslame S, Masseret E, Malledant Y, Launey Y, Seguin P. Low interleukin-10 release after ex vivo stimulation of whole blood is associated with persistent organ dysfunction in sepsis: A prospective observational study. Anaesth Crit Care Pain Med. 2019 Oct;38(5):485-491. doi: 10.1016/j.accpm.2019.01.009. Epub 2019 Feb 21. PMID 30797048
- [Background] Ikeda M, Matsumoto H, Ogura H, Hirose T, Shimizu K, Yamamoto K, Maruyama I, Shimazu T. Circulating syndecan-1 predicts the development of disseminated intravascular coagulation in patients with sepsis. J Crit Care. 2018 Feb;43:48-53. doi: 10.1016/j.jcrc.2017.07.049. Epub 2017 Jul 28. PMID 28843664
- [Background] Kjaergaard AG, Dige A, Nielsen JS, Tonnesen E, Krog J. The use of the soluble adhesion molecules sE-selectin, sICAM-1, sVCAM-1, sPECAM-1 and their ligands CD11a and CD49d as diagnostic and prognostic biomarkers in septic and critically ill non-septic ICU patients. APMIS. 2016 Oct;124(10):846-55. doi: 10.1111/apm.12585. Epub 2016 Aug 19. PMID 27539881
- [Background] Schuetz P, Plebani M. Can biomarkers help us to better diagnose and manage sepsis? Diagnosis (Berl). 2015 Jun 1;2(2):81-87. doi: 10.1515/dx-2014-0073. PMID 29540028
- [Background] Milbrandt EB, Reade MC, Lee M, Shook SL, Angus DC, Kong L, Carter M, Yealy DM, Kellum JA; GenIMS Investigators. Prevalence and significance of coagulation abnormalities in community-acquired pneumonia. Mol Med. 2009 Nov-Dec;15(11-12):438-45. doi: 10.2119/molmed.2009.00091. Epub 2009 Sep 8. PMID 19753144
- [Background] Beloncle F, Rousseau N, Hamel JF, Donzeau A, Foucher AL, Custaud MA, Asfar P, Robert R, Lerolle N. Determinants of Doppler-based renal resistive index in patients with septic shock: impact of hemodynamic parameters, acute kidney injury and predisposing factors. Ann Intensive Care. 2019 Apr 24;9(1):51. doi: 10.1186/s13613-019-0525-8. PMID 31020427
- [Background] Annane D, Ouanes-Besbes L, de Backer D, DU B, Gordon AC, Hernandez G, Olsen KM, Osborn TM, Peake S, Russell JA, Cavazzoni SZ. A global perspective on vasoactive agents in shock. Intensive Care Med. 2018 Jun;44(6):833-846. doi: 10.1007/s00134-018-5242-5. Epub 2018 Jun 4. PMID 29868972